CLINICAL TRIAL: NCT01723280
Title: Perioperative Inspiratory Oxygen Fraction - Effect on Occurrence of Subsequent Cancer After Abdominal Surgery (Follow-up of the PROXI Trial)
Brief Title: Supplemental Oxygen - Effect on Occurrence of Subsequent Cancer After Abdominal Surgery (Follow-up of the PROXI Trial)
Acronym: PROXI
Status: Completed | Type: Observational
Sponsor: Lars S. Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Lars S. Rasmussen, Professor, MD, PhD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: 2006-001710-32-follow-up; GCP-2006-101 (Other: Danish GCP-unit); KF 02 306766 (Other: Ethics committee)
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Laparotomy
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 80% oxygen group
  Interventions: Drug: Oxygen
- 30% oxygen group
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — During and 2 hrs after surgery

SUMMARY:
Aim: to investigate the effect of a high inspiratory oxygen fraction (FiO2) given during and after laparotomy procedures on occurrence of a subsequent, new or recurrent, cancer diagnosis at a long-term follow-up.

Background: A high inspiratory oxygen fraction (FiO2 = 0.80) has been linked to prevention of surgical site infection, but the Danish randomized clinical multicenter trial, the PROXI trial, found no difference in frequency of surgical site infection. In fact, long-term mortality was significantly increased with a hazards ratio of 1.30 in patients receiving 80% oxygen, and this appeared to be statistically significant in patients undergoing cancer surgery, but not in non-cancer patients.

At this point, no convincing mechanism explains the observed increased mortality after hyperoxia, as the long-term pathophysiological effects of oxygen are not fully understood.

Primary hypothesis of this follow-up study of the PROXI trial: Use of 80% oxygen increase the frequency of patients with a subsequent, new or recurrent, cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Laparotomy, acute or elective. In case of gynaecological surgery only if malignancy is suspected (defined as risk of ovarian malignancy index >200 or a specimen with atypical or neoplastic cells).

Exclusion Criteria:

* Other surgery within 30 days (except surgery in local anaesthesia).
* Chemotherapy within 3 months.
* Inability to give informed consent.
* Inability to keep oxygen saturation above 90% without supplemental oxygen (measured preoperatively by pulse oximetry).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the PROXI trial
Sampling Method: Non-Probability Sample
Enrollment: 1386 (Actual)
Dates: Start 2006-10; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with the composite outcome measure of either a subsequent, new or recurrent, cancer registration or a new histological specimen showing any neoplasm | 36-60 months after randomization

SECONDARY OUTCOMES:
Frequency of patients with subsequent, new or recurrent, cancer registration at the Danish Cancer Registry | 15-39 months after randomization
Frequency of patients with new histological specimen in the Danish Patobank showing any neoplasm | 36-60 months after randomization
Frequency of patients with new histological specimen in the Danish Patobank showing neoplasm of a histological type not previously diagnosed | 36-60 months after randomization
Frequency of patients with cancer as diagnosis code at a readmission | 36-60 months after randomization
Frequency of patients with cancer as primary diagnosis code at a readmission | 36-60 months after randomization
Duration of cancer-free survival, as assessed by Kaplan-Meier statistics | 36-60 months after randomization

OTHER OUTCOMES:
Type of new cancer registration | 15-39 months after randomization
Histological type of new cancer specimen | 36-60 months after randomization
Cause of death | 15-39 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. of Anesthesia, HOC, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Simonsen I, Pulawska T, Walker LR, Skovgaard N, Helto K, Gocht-Jensen P, Carlsson PS, Rask H, Karim S, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Perioperative oxygen fraction - effect on surgical site infection and pulmonary complications after abdominal surgery: a randomized clinical trial. Rationale and design of the PROXI-Trial. Trials. 2008 Oct 22;9:58. doi: 10.1186/1745-6215-9-58. PMID 18945347
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Hogdall C, Lundvall L, Svendsen PE, Mollerup H, Lunn TH, Simonsen I, Martinsen KR, Pulawska T, Bundgaard L, Bugge L, Hansen EG, Riber C, Gocht-Jensen P, Walker LR, Bendtsen A, Johansson G, Skovgaard N, Helto K, Poukinski A, Korshin A, Walli A, Bulut M, Carlsson PS, Rodt SA, Lundbech LB, Rask H, Buch N, Perdawid SK, Reza J, Jensen KV, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. JAMA. 2009 Oct 14;302(14):1543-50. doi: 10.1001/jama.2009.1452. PMID 19826023
- [Derived] Meyhoff CS, Jorgensen LN, Wetterslev J, Siersma VD, Rasmussen LS; PROXI Trial Group. Risk of new or recurrent cancer after a high perioperative inspiratory oxygen fraction during abdominal surgery. Br J Anaesth. 2014 Jul;113 Suppl 1:i74-i81. doi: 10.1093/bja/aeu110. Epub 2014 May 23. PMID 24860156